CLINICAL TRIAL: NCT05221255
Title: Effect of Spinal Magnetic Stimulation on Management of Functional Constipation in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Nehad Mohamed Elshatby Mahmoud, Physician, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0305398
Record Dates: First submitted 2022-01-10; First posted 2022-02-02 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Functional Constipation
Keywords: spinal magnetic stimulation, constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: interventional prospective trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Therapy (Sham Comparator): Patients will receive 12 sessions of biofeedback-assisted pelvic floor muscle relaxation plus non-real magnetic stimulation.
  Interventions: Other: spinal magnetic stimulation
- Spinal magnetic stimulation (Experimental): Patients will receive 12 sessions of biofeedback-assisted pelvic floor muscle relaxation followed by real spinal magnetic stimulation.
  Interventions: Other: spinal magnetic stimulation

INTERVENTIONS:
Other: spinal magnetic stimulation — * Biofeedback pelvic floor muscle training sessions will be performed for both groups for a total of 12 sessions. Menstruating women will be temporarily withdrawn from BF sessions till end of the menses. The session will last for 30 minutes of transrectal pressure biofeedback relaxation technique. Auditory and visual feedback will be provided in addition to positive verbal reinforcement.
  * Sham SMS will be used in the Sham group using the placebo program in the magnetic stimulation machine.
  * Spinal magnetic stimulation using the Neuro-MS/D machine. It will be used in spinal magnetic stimulation group, circular coil will be used to stimulate S2,3 and 4 sacral roots. Intensities will be adjusted to 50-70 % of maximal output (2.2 Tesla), stimulation frequency will be fixed at 20 Hz, burst length = 5 seconds, inter-burst interval = 25 seconds.

SUMMARY:
conservative management of functional constipation is a preferable method including biofeedback and spinal magnetic stimulation sessions

DETAILED DESCRIPTION:
Constipation varies in presentation and severity among patients and affects patients' quality of life of varied degrees depending on how it manifests and how severe it is. The prevalence of constipation in the general population is estimated to affect about 20% of the population

Spinal Magnetic Stimulation (SMS) is a non-invasive, painless neurophysiological treatment that uses extracorporeal magnetic stimulation to direct extracorporeal magnetic stimulation to the spinal nerves and deep muscles to aid bowl evacuation without the use of surgery. This noninvasive approach was created to help with micturition, expiration, and bowel function

The aim of this work is to study the efficacy of SMS and biofeedback versus biofeedback in the management of functional constipation.

ELIGIBILITY:
Inclusion Criteria:

* adults patients diagnosed by Rome IV criteria as having functional constipation

Exclusion Criteria:

* Patients younger than 18 years old.
* Patients with irritable bowel syndrome.
* Anal hemorrhoids or bleeding.
* Any condition that may complicate bowel problems, such as Parkinson's disease, stroke, or traumatic brain injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Number of weekly bowel movement | after 15 days
  Mean weekly complete spontaneous bowel movements.
The Bristol Stool Scale (from 1 to 5) | After 15 days
  Stool consistency
Numerical rating scale (from 0 to 10) | After 15 days
  pain assessment, zero indicates no pain, 10 indicates maximum pain degree
Patient Assessment of Constipation Quality of Life questionnaire | After 15 days
  Assessment of quality of life (from 9 to 127) lower scores indicating fewer problems
pressure manometry | After 15 days
  Assessment of pelvic floor power of contraction

SECONDARY OUTCOMES:
Number of weekly bowel movement | after one month
  Mean weekly complete spontaneous bowel movements.
The Bristol Stool Scale (from 1 to 5) | After one month
  Stool consistency
Numerical rating scale (from 0 to 10) | After one month
  pain assessment, zero indicates no pain, 10 indicates maximum pain degree
Patient Assessment of Constipation Quality of Life questionnaire | After one month
  Assessment of quality of life (from 9 to 127) lower scores indicating fewer problems
Pressure manometry | After one month
  Assessment of pelvic floor power of contraction

CONTACTS AND LOCATIONS:
Overall Officials: Nehad ElShatby, MD,PhD, Principal Investigator — Alexandria University
Locations (1):
- Nehad ElShatby, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be available with the corresponding author for three years after publishing the study, and ready to be shared with other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: from date of publication and 3 years after
Access Criteria: Contact the corresponding author via dr.nehad@yahoo.com